CLINICAL TRIAL: NCT01046032
Title: Metformin Treatment Before IVF in Women With Ultrasound Evidence of Polycystic Ovaries; a Prospective, Randomised, Double Blind, Placebo Study
Brief Title: Metformin Treatment Before in Vitro Fertilization (IVF) in Women With Ultrasound Evidence of Polycystic Ovaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Imperial College London (Other); University of Nottingham (Other)
Responsible Party: Mr Tim Child/Consultant Gynaecologist and Chief Investigator, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05/Q1605/87
Record Dates: First submitted 2010-01-03; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovaries; Ovarian stimulation; IVF; Ovarian hyperstimulation; Metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Drug (including placebo)
  Interventions: Drug: Metformin
- Sugar pill (Placebo Comparator): Drug (including placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Women were randomised to receive either metformin or placebo starting three weeks before initiation of a GnRH agonist during an IVF treatment cycle (seven weeks prior to oocyte collection and then stopped at oocyte collection). Seventy identical packs of metformin and 70 identical packs of placebo were supplied by DHP Ltd, Crickhowell, Powys (UK) a commercial clinical trial supplier. The randomisation service was provided by DHP Ltd.
  Arms: Metformin
Drug: Placebo — Women were randomised to receive either metformin or placebo starting three weeks before initiation of a GnRH agonist during an IVF treatment cycle (seven weeks prior to oocyte collection and then stopped at oocyte collection). Seventy identical packs of metformin and 70 identical packs of placebo were supplied by DHP Ltd, Crickhowell, Powys (UK) a commercial clinical trial supplier. The randomisation service was provided by DHP Ltd.
  Arms: Sugar pill

SUMMARY:
The aim of study was to investigate whether pre-treatment with metformin before and during IVF increases the live birth rate compared to placebo in women with sonographic evidence of polycystic ovaries (PCO), but without any clinical manifestations of polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

* Women attending with ovulatory PCO due to undergo IVF/ICSI treatment.
* First or second cycle of IVF/ICSI.
* If previously on metformin, a minimum one month washout period was required.
* Polycystic ovaries diagnosed by ultrasound presence of ≥12 follicles measuring 2-9 mm in diameter in at least one ovary and/or increased ovarian volume (≥10 ml).
* Written informed consent.

Exclusion Criteria:

* Clinical manifestations of PCOS, including any of the following:

  1. Oligo- or amenorrhoea with cycles ≥42 days apart.
  2. Anovulation with mid-luteal progesterone <16 nmol/L.
  3. Biochemical hyperandrogenism with serum testosterone ≥3.5 nmol/L and/or free androgen index >5 (FAI = [total testosterone/SHBG] x 100).
  4. Clinical hyperandrogenism with hirsutism or acne requiring treatment at least weekly.
* Age >38 years.
* BMI >35 kg/m2.
* Basal FSH >12 IU/L.
* Liver disease or ALT >80 IU/L.
* Renal disease, or creatinine >130 nmol/L.
* Alcoholism or drug abuse.
* Diabetes mellitus (evaluated by fasting glucose >6.7mmol/L).
* Per oral steroid treatment in last month.
* Cimetidine, anticoagulation, erythromycin, or other macrolides in last month.
* Hyperprolactinemia (Prolactin >700 mIU/L).
* Abnormal thyroid function tests (TSH outside of laboratory normal range).
* Congenital adrenal hyperplasia.

Max Age: 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Live birth rate | End of pregnancy

SECONDARY OUTCOMES:
Severe ovarian hyperstimulation syndrome | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Child, MA MD MRCOG, Study Director — University of Oxford; Alexander G Swanton, MBBS MRCOG, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - IVF Hammersmith, London
  - Nuture IVF Unit, Nottingham
  - Oxford Fertility Unit, Oxford

REFERENCES:
- [Background] Tang T, Glanville J, Orsi N, Barth JH, Balen AH. The use of metformin for women with PCOS undergoing IVF treatment. Hum Reprod. 2006 Jun;21(6):1416-25. doi: 10.1093/humrep/del025. Epub 2006 Feb 24. PMID 16501038
- [Background] Kjotrod SB, von During V, Carlsen SM. Metformin treatment before IVF/ICSI in women with polycystic ovary syndrome; a prospective, randomized, double blind study. Hum Reprod. 2004 Jun;19(6):1315-22. doi: 10.1093/humrep/deh248. Epub 2004 Apr 29. PMID 15117902
- [Derived] Swanton A, Lighten A, Granne I, McVeigh E, Lavery S, Trew G, Talmor A, Raine-Fenning N, Jayaprakasan K, Child T. Do women with ovaries of polycystic morphology without any other features of PCOS benefit from short-term metformin co-treatment during IVF? A double-blind, placebo-controlled, randomized trial. Hum Reprod. 2011 Aug;26(8):2178-84. doi: 10.1093/humrep/der120. Epub 2011 May 18. PMID 21593045